CLINICAL TRIAL: NCT05436236
Title: Cannabis Consumption Effect on Gastric Volumes
Brief Title: Effect of Cannabis (Marijuana) on Stomach Emptying Before Surgery
Status: Withdrawn | Type: Observational
Why Stopped: Investigator decision
Sponsor: The Guthrie Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 2204-15
Record Dates: First submitted 2022-06-23; First posted 2022-06-29 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Gastric Emptying; Cannabis
MeSH Terms: conditions — Marijuana Abuse

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: People who self-report that they do not use cannabis.
- Cannabis: People who self-report that they use cannabis.

SUMMARY:
The purpose of this research is to study the effect of cannabis (marijuana) on gastric (stomach) emptying before surgery. The study will include people who use cannabis (study group) and people who do not use cannabis (control group).

DETAILED DESCRIPTION:
About 108 people will take part in this study (54 in the study group and 54 in the control group). Subjects will have an ultrasound of the abdomen before their scheduled surgery. The ultrasound will determine how much fluid remains in the abdomen.

Researchers will also review subjects' medical records and will include: age, body mass index, history of cannabis use including how often and how consumed, reason for surgery, and length of time without eating before surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18 years and older
* Planned surgery at one of two hospitals within the healthcare system
* Willing to state if they use or do not use cannabis
* Able to read and consent on their own behalf

Exclusion Criteria:

* Cognitively impaired
* Unable to read
* Children under the age of 18
* Pregnant women - Pregnancy status will be obtained from the routine pregnancy test performed prior to surgery
* History of gastroparesis
* Gastric surgeries
* Advanced liver or renal dysfunction
* Critically ill
* Emergent/urgent cases

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects 18 years and older with a planned surgery at one of two hospitals within the healthcare system, who are willing to state if they use or do not use cannabis
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Gastric content volume | pre-operative
  Gastric content volume as assessed by ultrasound prior to surgery

SECONDARY OUTCOMES:
Frequency of cannabis use | 3 months prior to surgery
  number of times per week patient uses cannabis
Cannabis use (chronic yes or no) | 1 year prior to surgery
  Yes or No for chronic cannabis use
Route of cannabis consumption | 3 months prior to surgery
  Categories of how cannabis is consumed (smoke, vape, other)
Time since last food; Nil per os (NPO) time | 24 hours prior to surgery
  Length of time patient had no food prior to surgery

CONTACTS AND LOCATIONS:
Overall Officials: Neel Kapoor, DO, Principal Investigator — The Guthrie Clinic

IPD SHARING:
Plan to Share IPD: No